CLINICAL TRIAL: NCT01624545
Title: To Scan or Not to Scan: The Role of Follow-up CT Scanning for Management of Chronic Subdural Hematoma After Neurosurgical Evacuation - a Prospective, Randomized, Controlled Trial
Brief Title: To Scan or Not to Scan: The Role of Follow-up CT Scanning for Management of Chronic Subdural Hematoma After Neurosurgical Evacuation
Acronym: TOSCAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 218/10; 2179
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Chronic Subdural Hematoma
Keywords: chronic subdural hematoma; burr hole trepanation; radiologic follow-up; outcome; recurrence
MeSH Terms: conditions — Hematoma, Subdural, Chronic; Recurrence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Patients in this study arm will receive a cranial CT scan on day 2 and day 30 after evacuation of a chronic subdural hematoma in addition to neurological evaluation on day 2 and 30.
  Interventions: Other: cranial CT scan
- 2 (No Intervention): Patients in this study arm will undergo neurological evaluation on day 2 and day 30 without follow-up CT scan.

INTERVENTIONS:
Other: cranial CT scan — Patients in this study arm will receive a cranial CT scan on day 2 and day 30 after evacuation of a chronic subdural hematoma in addition to neurological evaluation on day 2 and 30.
  Arms: 1

SUMMARY:
Chronic subdural hematoma (CSH) is one of the most common bleedings of the head. These hematomas develop after minor head trauma and increase in size over weeks. Patients usually present with headaches, gait disturbances, language problems or confusion. The state of the art treatment of a symptomatic chronic subdural hematoma is to remove the hematoma by burr hole trepanation.

The optimal follow-up for operated patients remains controversial. Due to the known high rate of a second hematoma at the same place (usually within weeks), one strategy is to perform serial computer tomography scans in order to identify recurrent hematomas early. The radiologic evidence of a second hematoma often leads to reoperation, even if the patient has no, or just slight symptoms. Another strategy after surgical hematoma evacuation is to closely follow the patient with neurological examinations and perform neuroimaging only in case of new symptoms. Advocators of this strategy argue that a follow-up with routine CT scans may be harmful due to additional and maybe unnecessary surgeries and hospital days in a patient population marked by advanced age and fragility.

The aim of the current study is to evaluate the role of computer tomography scanning in the postoperative follow-up after removal of a chronic subdural hematoma. Participants of this study will be allocated by chance to one of two study groups: Patients allocated to group A will receive a computer tomography scan on day 2 and again on day 30 after surgery in addition to a clinical examination. Patients allocated to group B will be examined clinically on day 2 and day 30 without computer tomography. All patients will undergo a final clinical examination after 6 months. The study will recruit 400 patients.

DETAILED DESCRIPTION:
Background

Chronic subdural hematoma (CSH) is one of the most common intracranial bleedings in patients over 60 years of age and a frequently found neurosurgical entity. Age related brain atrophy leads to enlargement of the subarachnoid space, a space limited by the dura mater and the arachnoid membrane. Blood vessels that occupy this space are being stretched and may rupture after a minor head trauma. Although the resulting bleeding itself is often without noticeable consequence for the patient, the anatomical outcome may be serious as it enlarges the subdural space. The formation of new leaky capillary-like vessels and/or volume enhancing osmotic gradients lead to the enlargement of the subdural hematoma over weeks, filling the intracranial space and compressing the brain. Headaches, gait disturbances, language problems, hemiparesis and decreased consciousness are among the many presenting symptoms and tend to develop over days or weeks.

Computed tomography (CT) scan or magnetic resonance imaging (MRI) of the head typically reveals the blood accumulation in the subdural space. Standard treatment includes the evacuation of the subdural blood through burr holes (see below) under either local or general anesthesia. In cases when a hematoma clot cannot be evacuated through burr holes a small craniotomy is performed. CSH is feared for its high recurrence rate (between 9 and 27%) that mostly occurs within 3 months of the initial operation.

The optimal follow-up course for operated patients remains controversial. Due to the high rate of recurrences, one strategy is to perform serial CT scans in order to identify recurrent hematomas early. The radiologic evidence of a recurrent or significant persistent hematoma often leads to reoperation. Another strategy after surgical hematoma evacuation is to closely follow the patient with neurological examinations and perform neuroimaging only in case of persistent or new neurologic deficits. Advocators of this strategy argue that follow up with routine CT scans may be harmful due to additional and maybe unnecessary surgeries and hospital days in a patient population marked by advanced age and fragility.

However, even when neuroimaging is done routinely, no correlation has been observed between the radiologic evidence of a hematoma remnant and the reoperation rate. This observation has been reported by Mori and Maeda in a retrospective analysis of 500 patients. Some persistent hematoma is almost always seen after the surgical intervention and there seems to be a correlation between the re-expansion rate of the brain and the likelihood of hematoma recurrence. However, the correlation is weak and of little practical value for patient treatment. The high incidence of hematoma remnants in post-op imaging complicates the indication for re-operation of a recurrent CSH solely by imaging criteria. Since the presence and the amount of remnant hematoma after the operation is a poor predictor of future recurrent hematoma some clinicians refrain from postoperative CT scans and rely solely on neurological assessments. If patients become symptomatic, serial CT scans are performed and surgery is scheduled in cases of persistent, enlarging or new hematoma. The discrepancy in follow-up strategy reflects our current incomplete understanding of the pathophysiology of CSH and its recurrence.

The aim of the current study is to evaluate the role of CT scanning in the postoperative treatment course after neurosurgical evacuation of CSH in a prospective, randomized controlled trial.

Objective

The hypothesis of interest to test in this trial is that a follow-up protocol without any CT scan is not inferior to a follow-up protocol with serial CT scans after neurosurgical evacuation of CSH as assessed with the modified Rankin scale at 6 months. Additional hypotheses of interest are that the size/volume/features of the hematoma rest/remnant in an early (<72 hours) CT scan after neurosurgical evacuation is not correlated to the neurological status of the patient and that the size/volume/features of the hematoma rest/remnant on post-op CT scans is not predictive for reoperation.

Methods

Patients will be screened and included into this study within 48 hours after surgery for a chronic subdural hematoma (burr hole trepanation and insertion of drainage). Study patients are randomized (1:1) on day 2 after surgery into CT-Scan arm (group A) or Clinical arm (group B). A CT scan is scheduled for patients of group A on day 2 and 30 after surgery. Patients of both study groups (A and B) will receive a neurological follow-up examination at day 2, 30 days and 6 months after surgery. Regardless of randomization all patients will receive CT scanning if judged necessary on clinical grounds at any time.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed chronic subdural hematoma by CT scan or MRI, operated within the last 48 hours
* Age 18 years or older
* Written informed consent from the patient to participate in the study

Exclusion Criteria

* Moribund state of health prohibiting surgery
* Foreseeable difficulties in follow-up due to geographic reasons (e.g. patients living abroad)
* Recurrent hematoma if the first surgery was performed before study start
* CSH due to spontaneous spinal CSF fistula or meningeosis carcinomatosa
* Pregnancy
* Patient with Metastatic Disease and a high possibility to pass away in the next 6 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2017-02-06 (Actual); Study Completion 2017-02-06 (Actual)

PRIMARY OUTCOMES:
modified Rankin Scale | 6 months

SECONDARY OUTCOMES:
Rate of reoperation | 6 months
Mini Mental Status | 6 months
NIHSS | 6 months
QLQ-C30 | 6 months
Total length of hospitalisation | 6 months
Influence of the size and radiological features of the hematoma on rate of recurrence | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Philippe E Schucht, MD, Principal Investigator — Inselspital Bern, University Bern
Locations (1):
- Department of Neurosurgery, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Background] Mori K, Maeda M. Surgical treatment of chronic subdural hematoma in 500 consecutive cases: clinical characteristics, surgical outcome, complications, and recurrence rate. Neurol Med Chir (Tokyo). 2001 Aug;41(8):371-81. doi: 10.2176/nmc.41.371. PMID 11561347
- [Background] Torihashi K, Sadamasa N, Yoshida K, Narumi O, Chin M, Yamagata S. Independent predictors for recurrence of chronic subdural hematoma: a review of 343 consecutive surgical cases. Neurosurgery. 2008 Dec;63(6):1125-9; discussion 1129. doi: 10.1227/01.NEU.0000335782.60059.17. PMID 19008766
- [Background] Forster MT, Mathe AK, Senft C, Scharrer I, Seifert V, Gerlach R. The influence of preoperative anticoagulation on outcome and quality of life after surgical treatment of chronic subdural hematoma. J Clin Neurosci. 2010 Aug;17(8):975-9. doi: 10.1016/j.jocn.2009.11.023. Epub 2010 May 23. PMID 20580997
- [Background] Abouzari M, Rashidi A, Rezaii J, Esfandiari K, Asadollahi M, Aleali H, Abdollahzadeh M. The role of postoperative patient posture in the recurrence of traumatic chronic subdural hematoma after burr-hole surgery. Neurosurgery. 2007 Oct;61(4):794-7; discussion 797. doi: 10.1227/01.NEU.0000298908.94129.67. PMID 17986941
- [Background] Oishi M, Toyama M, Tamatani S, Kitazawa T, Saito M. Clinical factors of recurrent chronic subdural hematoma. Neurol Med Chir (Tokyo). 2001 Aug;41(8):382-6. doi: 10.2176/nmc.41.382. PMID 11561348
- [Background] Santarius T, Kirkpatrick PJ, Ganesan D, Chia HL, Jalloh I, Smielewski P, Richards HK, Marcus H, Parker RA, Price SJ, Kirollos RW, Pickard JD, Hutchinson PJ. Use of drains versus no drains after burr-hole evacuation of chronic subdural haematoma: a randomised controlled trial. Lancet. 2009 Sep 26;374(9695):1067-73. doi: 10.1016/S0140-6736(09)61115-6. PMID 19782872
- [Background] Lee HY, Ju YM, Lee MH, Lee SJ, Chang WH, Imm CW. A case of post-traumatic coronary occlusion. Korean J Intern Med. 1991 Jan;6(1):33-7. doi: 10.3904/kjim.1991.6.1.33. PMID 1742254